CLINICAL TRIAL: NCT00126828
Title: A Phase I/II Study of Radiation Dose Intensity Concurrent With Chemotherapy For Limited Stage Small Cell Lung Cancer
Brief Title: Study of Radiation Dose Intensity Concurrent With Chemotherapy For Limited Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LU-11-0031 / 17141; PCRP-07
Record Dates: First submitted 2005-08-03; First posted 2005-08-05 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2011-10

CONDITIONS: Carcinoma, Small Cell
Keywords: radiotherapy, conformal; lung neoplasm; radiotherapy dosage
MeSH Terms: conditions — Carcinoma, Small Cell; Lung Neoplasms

INTERVENTIONS:
Procedure: External beam radiotherapy

SUMMARY:
Patients who have limited stage small cell lung cancer are presently treated with chemotherapy and radiation therapy (RT). Despite this aggressive treatment the vast majority of patients will have their cancer recur after treatment. A recurrence is not curable at this time, therefore efforts to reduce recurrence rates are desirable. Due to the sensitivity of surrounding structures in the chest to radiation, it has not been possible to give doses that can cure most tumours. Three-dimensional conformal radiotherapy is a special form of radiation therapy that allows doctors to reduce the amount of radiation dose to normal tissues and therefore reduce toxicity and in turn, let them safely increase the dose to tumours. The purpose of this study is to determine whether the combination of three-dimensional conformal radiotherapy and chemotherapy will be a more effective treatment. If the treatment is found to be safe for the first group of patients, then the total radiation dose will be increased for the next group of patients who are treated on this study.

DETAILED DESCRIPTION:
Radiotherapy represents one of the primary treatment modalities for patients with limited stage small cell lung cancer (SCLC). With contemporary concurrent radiotherapy and chemotherapy, approximately 20% of patients survive 5 years. While distant metastases are common, local (intrathoracic) failures are common as well, occurring in 40% of treated patients. Reducing local failure rates may lead to improved survival for these patients. There appears a growing body of data, which suggests a radiation dose response relationship for SCLC. However, the close proximity of critical normal structures, such as the spinal cord and esophagus, to the primary tumour limits the prescription dose in conventional radiotherapy. Three Dimensional Conformal Radiotherapy (3DCRT) offers the possibility of reducing normal tissue irradiation and hence reducing the treatment toxicity while maintaining the dose of radiation to the tumour. Another strategy is accelerated fractionation, which shortens the treatment time by allowing less opportunity for tumour cell repopulation. The use of 3DCRT with larger radiation fraction size should maintain satisfactory treatment related toxicity while permitting the potential gains of accelerated fractionation and dose escalation. In this study, patients with limited stage SCLC who are eligible will be treated with a large field (low dose) radiotherapy followed by accelerated 3DCRT given concurrently with standard Cisplatin Etoposide chemotherapy.

Primary Objective: To determine the maximum tolerable dose of radiotherapy for SCLC

Secondary Objectives:

1. To assess treatment toxicity
2. To assess quality of life and retention of pulmonary function
3. To assess progression-free survival on this regimen

Schema: Eligible patients will receive 4 cycles of Cisplatin Etoposide chemotherapy. Thoracic radiotherapy will be given concurrently starting with cycle #2 of chemotherapy. Only one dose level will be open at a time. Four dose levels are planned all delivered in 25 fractions once daily over 5 weeks:

1. 50 Gy (2 Gy per fraction),
2. 58 Gy,
3. 62 Gy,
4. 65 Gy. Patients, who achieve a complete response at the end of chemotherapy and thoracic radiotherapy, will receive prophylactic cranial irradiation.

Evaluation and Follow-up: Patients will be assessed and evaluated at least weekly during radiation therapy. Following treatment, patients will be seen 1 month after the completion of treatment, then every 3 months until 2 years, then every 6 months. Chest x-rays will be performed at each follow-up. CT scan of chest and pulmonary function tests will be performed every 6 months for the first 2 years, then yearly.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven small cell lung cancer
* Age equal to or greater than 18 years
* Good performance status
* Signed study consent form

Exclusion Criteria:

* Patients who have undergone resection
* Wrong histology
* Previous thoracic/neck radiotherapy
* Prior chemotherapy
* Previous ME within 6 months
* Pregnant
* Tumour too large to irradiate safely

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18
Dates: Start 2003-01; Primary Completion 2007-09 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
grade 3 RT toxicity rate

SECONDARY OUTCOMES:
disease free
overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Peter Venner, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada